CLINICAL TRIAL: NCT02603887
Title: Pilot Single Arm, Single Center, Open Label Trial of Pembrolizumab in Patients With Intermediate and High Risk Smoldering Multiple Myeloma
Brief Title: Pembrolizumab in Treating Patients With Intermediate or High-Risk Smoldering Multiple Myeloma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0371; NCI-2015-02135 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0371 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Smoldering Plasma Cell Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This pilot early phase I trial studies pembrolizumab in treating patients with slow growing (smoldering) multiple myeloma with intermediate or high-risk of spreading. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall response rate after 8 cycles of treatment according to the International Myeloma Working Group Criteria (IMWG).

SECONDARY OBJECTIVES:

I. To determine time to progression to multiple myeloma (TTP) at 30 months from study entry.

II. To determine overall survival (OS). III. To determine duration of response (DOR). IV. To determine the clinical benefit rate (CBR) after 8 cycles of treatment according to the modified IMWG Criteria for multiple myeloma (MM).

V. To evaluate safety and tolerability of single agent treatment in this population.

EXPLORATORY OBJECTIVES:

I. Rate of minimal residual disease (MRD) negativity at complete remission (CR).

II. Molecular profiling (including whole exome sequencing and gene expression profiling) and cellular (including flow cytometry) profiling at baseline and/or at progression using bone marrow aspirate samples and peripheral blood.

III. Immunophenotypic characterization of dendritic, T-, B-, natural killer (NK)- and natural killer T (NKT)-cells, and inhibitory/activation markers on tumor cells at baseline and at completion of 8 cycles of therapy in bone marrow aspirate samples and/or peripheral blood.

IV. Evaluation of changes in PD-L1 and PD-1 expression at baseline/end of 8 cycles of treatment and correlate with clinical response.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with intermediate or high-risk smoldering multiple myeloma (SMM) are eligible; patients need to have clonal bone marrow plasma cells >= 10% and/or monoclonal spike in blood of >= 3 g/dL and/or monoclonal urine component (Bence jones proteinuria) >= 500 mg/24 hours and need to meet subject inclusion criteria and exclusion criteria as per below
* Patients must have histologically confirmed SMM based on the following criteria:

  * (A) Mayo clinic criteria (patient must have at least 2 risk factors present):

    * 1. Bone marrow core biopsy plasma cell involvement by cluster of differentiation (CD)138 immunohistochemistry >= 10%
    * 2. Monoclonal spike >= 3 g/dL
    * 3. Free light chain ratio in serum < 0.125 or > 8; *2 of 3 risk factors: intermediate risk for progression at a rate of 51% at 5 years, *3 of 3 risk factors: high risk for progression at a rate of 76% at 5 years
  * OR (B) Programa para el Tratamiento de Hemopatias Malignas (PETHEMA) criteria (patient must have at least 1 risk factor present)

    * 1. >= 95% abnormal plasma cells/total plasma cells in bone marrow compartment
    * 2. Immunoparesis *1 of 2 risk factors: intermediate risk for progression at a rate of 46% at 5 years, *2 of 2 risk factors: high risk for progression at a rate of 72% at 5 years
  * OR (C) Southwestern Oncology Group (SWOG) criteria (patient must have 2 risk factors present or one risk factor if this risk factor is a 70-gene signature (GEP70) score of > 37.2)

    * 1. Monoclonal spike >= 3 g/dL
    * 2. Involved free light chain >= 25 mg/dL
    * 3. GEP70 risk score > 37.2 *>= 2 risk factors: high risk of progression at a rate of 70% at 2 years*; we would also include patients with 1 risk factor as long as this risk factor is GEP70 risk score > 37.2 since patients with this risk factor have an intermediate risk of progression at a rate of 50% at 2 years
* Creatinine clearance >= 50 ml/min; creatinine clearance (CrCl) will be calculated by Cockcroft-Gault method
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count (ANC) >= 1.0 x 10^9 /L
* Hemoglobin >= 10 g/dL
* Platelet count >= 50 x 10^9/L
* Bilirubin < 1.5 x the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3.0 x ULN
* Subjects must be able to give informed consent
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Evidence of myeloma defining events or biomarkers of malignancy due to underlying plasma cell proliferative disorder meeting at least one of the following

  * 1) Hypercalcemia: serum calcium > 0.25 mmol/L (> 1 mg/dL) higher than the upper limit of normal or > 2.75 mmol/L (> 11 mg/dL)
  * 2) Renal insufficiency: creatinine clearance < 40 ml/min or serum creatinine > 2 mg/dL
  * 3) Anemia: hemoglobin value < 10 g/dL or 2 g/dL < normal reference
  * 4) Bone lesions: one or more osteolytic lesions on skeletal radiography, computerized tomography (CT) or 2-deoxy-2[F-18] fluoro-D-glucose positron emission tomography CT (PET-CT)
  * 5) Clonal bone marrow plasma cell percentage >= 60%
  * 6) Involved: uninvolved serum free light chain ratio >= 100 measured by Freelite assay (The Binding Site Group, Birmingham, United Kingdom [UK])
  * 7) > 1 focal lesions on magnetic resonance imaging (MRI) studies (each focal lesion must be 5 mm or more in size), if clinically indicated
* Prior or concurrent systemic treatment for SMM; a) bisphosphonates are permitted; b) treatment with corticosteroids is not permitted; c) radiotherapy is not permitted; d) prior treatment for smoldering multiple myeloma with chemotherapy agents approved for the treatment of multiple myeloma is not permitted
* Plasma cell leukemia
* Pregnant or lactating females; breastfeeding should be discontinued if the mother is treated with pembrolizumab
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-programmed death ligand 2 (PD-L2) agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy; Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Evidence of interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Saini, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Manasanch EE, Han G, Mathur R, Qing Y, Zhang Z, Lee H, Weber DM, Amini B, Berkova Z, Eterovic K, Zhang S, Zhang J, Song X, Mao X, Morgan M, Feng L, Baladandayuthapani V, Futreal A, Wang L, Neelapu SS, Orlowski RZ. A pilot study of pembrolizumab in smoldering myeloma: report of the clinical, immune, and genomic analysis. Blood Adv. 2019 Aug 13;3(15):2400-2408. doi: 10.1182/bloodadvances.2019000300. PMID 31405950
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period was between July 2016 and August 2017
Pre-assignment Details: 20 participants were consented. 13 participants were treated at MD Anderson Cancer Center. An additional participant started stage 2 that did not participate in Stage 1"
Groups:
- Treatment (Pembrolizumab): Pembrolizumab 200 mg, 30 minute IV infusion every 21 days up to 24 cycles if equal or higher than minor response and without serious adverse events after 8 cycles
Period: Stage 1
Arm/Group | Treatment (Pembrolizumab)
Started | 12
Cycle 1 | 12
Cycle 8 | 7
Completed | 7
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Disease progression | 1
Period: Stage 2
Arm/Group | Treatment (Pembrolizumab)
Started | 1
Cycle 1 | 1
Cycle 8 | 0
Completed | 0
Not Completed | 1
Not completed — FDA guidance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [59 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Myeloma related labs [Median (Inter-Quartile Range); unit: gm/dL] — Measure Description: Laboratory exams including hemoglobin, calcium, creatinine, serum paraprotein, bence jones urine protein, kappa and lambda free light chain, free light chain ratio, involved:uninvolved ratio, B2 microglobulin, LDH and bone marrow biopsy plasma cell percentage, needed to assess properly a patient with plasma cell dyscrasia
  gm/dL
    Hemoglobin | 12.4 [11.95 to 13.95]
    Serum paraprotein | 1.9 [0.8 to 3.15]
Myeloma related labs [Median (Inter-Quartile Range); unit: mg/dL] — Measure Description: Laboratory exams including hemoglobin, calcium, creatinine, serum paraprotein, bence jones urine protein, kappa and lambda free light chain, free light chain ratio, involved:uninvolved ratio, B2 microglobulin, LDH and bone marrow biopsy plasma cell percentage, needed to assess properly a patient with plasma cell dyscrasia
  mg/dL
    Calcium | 9.3 [8.7 to 9.55]
    Creatinine | .88 [0.79 to 1.04]
Myeloma related labs [Median (Inter-Quartile Range); unit: mg/L] — Measure Description: Laboratory exams including hemoglobin, calcium, creatinine, serum paraprotein, bence jones urine protein, kappa and lambda free light chain, free light chain ratio, involved:uninvolved ratio, B2 microglobulin, LDH and bone marrow biopsy plasma cell percentage, needed to assess properly a patient with plasma cell dyscrasia
  mg/L
    B2 microglobulin | 1.9 [1.75 to 2.3]
    Kappa free light chain | 127.04 [18.18 to 277.48]
    Lambda free light chain | 8.08 [6.74 to 14.59]
Myeloma related lab Lactate dehydrogenase [Median (Inter-Quartile Range); unit: u/L] | 439 [349.5 to 488]
Myeloma related lab Bone marrow biopsy plasma cells [Median (Inter-Quartile Range); unit: percentage of plasma cells] | 30 [17.5 to 45]
Myeloma related lab Bence Jones urine protein [Median (Inter-Quartile Range); unit: mg/day] | 6 [0 to 30.5]
Myeloma related labs [Median (Inter-Quartile Range); unit: ratio] — Measure Description: Measure Description: Laboratory exams including hemoglobin, calcium, creatinine, serum paraprotein, bence jones urine protein, kappa and lambda free light chain, free light chain ratio, involved:uninvolved ratio, B2 microglobulin, LDH and bone marrow biopsy plasma cell percentage, needed to assess properly a patient with plasma cell dyscrasia
  ratio
    Free Light Chains (FLCs) ratio | 12.27 [2.44 to 38.25]
    Involved:Uninvolved ratio | 17.95 [6.44 to 38.25]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate is defined as patients who have achieved partial response or higher as described per IMWG criteria for multiple myeloma after 8 cycles of therapy with pembrolizumab. Will be measured according to International Myeloma Working Group Criteria (IMWG) criteria. Response rate will be estimated accordingly. Each cycle has a duration of 21 days.
Time Frame: From cycle 1 to cycle 8, up to 168 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 13
Participants | 1

2. Secondary Outcome: Number of Participants That Had Progression to Multiple Myeloma
Description: Progressive disease assessed by IMWG criteria for multiple myeloma after 8 cycles of therapy with pembrolizumab.
Time Frame: At 30 months from study entry
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 13
Participants | 3

3. Secondary Outcome: Clinical Benefit Rate
Description: Minor response or better assessed by IMWG criteria for multiple myeloma after 8 cycles of therapy with pembrolizumab
Time Frame: From cycle 1 to cycle 8, up to 168 days
Population: Clinical benefit rate is described as minor response or better assessed by IMWG criteria for multiple myeloma after 8 cycles of therapy with pembrolizumab. 1 participant of 13 achieved sCR
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 13
Participants | 1

4. Secondary Outcome: Overall Survival
Description: Participants in a study or treatment group who are still alive for a certain period of time after they were diagnosed with or started treatment for a disease
Time Frame: Time of start of treatment to death from any cause up to 2 years and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 13
Participants | 12

ADVERSE EVENTS:
Time Frame: From time the consent form is signed through 90 days following cessation of treatment and at each examination on the Adverse Event case report/forms/worksheet, up to 2 years and 6 months
Description: All adverse events were recorded on the adverse event case report/worksheet by the principal investigator and/or research team, as well as evaluated by a qualified physician
Groups:
- Single Arm, Intermediate-high Risk SMM Participants: Pembrolizumab 200 mg, 30 minute IV infusion every 21 days up to 24 cycles if equal or higher than minor response and without serious adverse events after 8 cycles
Arm/Group | Single Arm, Intermediate-high Risk SMM Participants
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm, Intermediate-high Risk SMM Participants (N=13)
Transaminitis (Hepatobiliary disorders) | 1 — All adverse events were recorded on the adverse event case report/worksheet by the principal investigator and/or research team, as well as evaluated by a qualified physician
Acute kidney injury (Renal and urinary disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm, Intermediate-high Risk SMM Participants (N=13)
Acute kidney injury (Renal and urinary disorders) | 2
Alanine aminotranferase increased (Blood and lymphatic system disorders) | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 5
Anorexia (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Autoimmune disorder (Immune system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Blurred vision (Eye disorders) | 1
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 1
Chills (General disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increased (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 6
Dizziness (Ear and labyrinth disorders) | 3
Dry eye (Eye disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Edema limbs (Skin and subcutaneous tissue disorders) | 4
Endocrine disorders - Other, specify (Endocrine disorders) | 3
Epistaxis (General disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Fatigue (General disorders) | 10
Fever (General disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (General disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hepatobiliary disorders - Other, specify (Gastrointestinal disorders) | 1
Hot flashes (General disorders) | 2
Hypercalcemia (Blood and lymphatic system disorders) | 1
Hyperglycemia (Blood and lymphatic system disorders) | 6
Hyperuricemia (Blood and lymphatic system disorders) | 1
Hypocalcemia (Blood and lymphatic system disorders) | 2
Hypomagnesemia (Blood and lymphatic system disorders) | 4
Hyponatremia (Blood and lymphatic system disorders) | 1
Hypophosphatemia (Blood and lymphatic system disorders) | 2
Insomnia (General disorders) | 2
Lipase increased (Blood and lymphatic system disorders) | 3
Memory impairment (General disorders) | 1
Metabolism and nutrition - Other, specify (Metabolism and nutrition disorders) | 4
Mucositis oral (General disorders) | 2
Muscoloeskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Neck edema (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Neoplasm benign, malignant and unspecified (incl cyst and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 1
Pain (General disorders) | 4
Palpitations (Cardiac disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Photophobia (Eye disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 1
Prostate infection (Infections and infestations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Serum amylase increased (Respiratory, thoracic and mediastinal disorders) | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3
Tinnutis (Ear and labyrinth disorders) | 1
Transaminitis (Hepatobiliary disorders) | 1
Tremor (Nervous system disorders) | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3
Urinary frequency (Renal and urinary disorders) | 2
Urinary tract infection (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Weight loss (Metabolism and nutrition disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT02603887/Prot_SAP_000.pdf